CLINICAL TRIAL: NCT06427161
Title: Dextrose Prolotherapy Versus Low Level Laser Therapy in Treatment of Patients With Obstructive Sleep Apnea Syndrome
Brief Title: Dextrose Prolotherapy Versus LLLT in Treatment of Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amira attia, Assistant professor of oral and maxillo-facial surgery Faculty of Dentistry, Mansoura University, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R.23.03.2095-2023/03/07
Record Dates: First submitted 2024-05-16; First posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Obstructive Sleep Apnea
Keywords: Dextrose; LLLT; obstructive sleep apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Glucose

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Ipatients were treated with LLLT. (Active Comparator): patients were treated with LLLT.
  Interventions: Procedure: LLLT application; Procedure: dextrose injection
- Group II (Active Comparator): patients were treated with dextrose injection.
  Interventions: Procedure: LLLT application; Procedure: dextrose injection

INTERVENTIONS:
Procedure: LLLT application — The LLLT group received the laser application at 8 points, once a week, over a 2-month period, totaling 8 sessions. Each point was stimulated for 8 seconds in the soft palate, uvula, pharyngeal walls, palatine tonsils, and on the tongue base. LLLT protocol: Diode laser 810nm in continuous contact mode was used, and the radiant energy was 2J (250uw X 8 sec) for each point. Total energy was 16J (2J X 8 points) for each session.
Procedure: dextrose injection — 25% dextrose was injected in the same 8 points; 1/2 ml for each point, total 4ml for each session. The injection was done weekly, up to 4 sessions.

SUMMARY:
This study was conducted on 26 patients with obstructive sleep apnea. The patients were divided randomly and equally into two equal groups. In group I, the patients were treated with LLLT, while in group II, the patients were treated with dextrose injection. The patients were evaluated by: Medical history utilizing sleep unit medical sheet, physical examination including: anthropometric measures, epworth sleepiness scale, and Berlin questioner, and Polysomnography

DETAILED DESCRIPTION:
This study was conducted on 26 patients with OSA attending to sleep disorders breathing Unit, Chest Department and oral and maxillofacial department at Mansoura University confirmed by polysomnography. The study was implemented over 2 months. The patients were divided randomly and equally into two therapy groups each compromise 13 patients:

Group I: patients will be treated with LLLT. Group II: patients will be treated with dextrose injection.

Interventions:

The LLLT group received the laser application at 8 points, once a week, over a 2-month period, totaling 8 sessions. Each point was stimulated for 8 seconds in the soft palate, uvula, pharyngeal walls, palatine tonsils, and on the tongue base. LLLT protocol: Diode laser 810nm in continuous contact mode will be used, and the radiant energy will be 2J (250uw X 8 sec) for each point. Total energy will be 16J (2J X 8 points) for each session.

Dextrose injection Protocol: 25% dextrose was injected in the same 8 points; 1/2 ml for each point, total 4ml for each session. The injection was done weekly, up to 4 sessions.

Clinical assessment

* Medical history utilizing sleep unit medical sheet will be taken from all patients: Attention was given to Night symptoms such as snoring, choking, witnessed apnea, bad dreams, and nocturia, and daytime symptoms (morning headache, excessive daytime sleepiness.
* Physical examination including: Anthropometric measures: Height, weight, body-mass index (BMI), teeth imprint, abdominal circumference, Epworth sleepiness scale (Arabic version), and Berlin questioner (Arabic version)
* Polysomnography

ELIGIBILITY:
Inclusion Criteria:

* All adult patients, diagnosed as having OSA after full night polysomnography. • BMI is between 28 kg/m2 and 40 kg/m2 at enrollment

Exclusion Criteria:

1. Pregnant patients
2. Active infectious disease (flu like symptoms).
3. Serious co-morbidity such as chronic or decompensated liver disease, and chronic kidney disease with creatinine clearance less than 30%.
4. Patients with neuromuscular disorders.
5. Previous trauma to the head, and neck.
6. Obvious fixed upper airway obstructions (tumors, polyps, nasal obstruction).
7. Tonsil size ≥ +3.
8. Clinical evidence of severe chronic obstructive or restrictive pulmonary disease (for example chronic bronchitis, emphysema, pulmonary fibrosis).
9. Active, severe pulmonary vascular disease (for example pulmonary arterial hypertension or pulmonary embolism).
10. Surgical resection for cancer or congenital malformations in the larynx, tongue, or throat (with exception of tonsillectomy and/or adenoidectomy).
11. History of radiation therapy to neck or upper respiratory tract
12. Patients with any cardiac diseases such as heart failure, rheumatic heart diseases, coronary artery disease, and myocardial infarction (MI).
13. Patients take up medications that will alter pain perception.
14. History of dementia or active psychiatric disease that may impact study compliance.
15. Patients who refuse the procedure.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-04-21 (Actual)

PRIMARY OUTCOMES:
Epworth sleepiness scale | 1 week after last treatment session.
  No chance of dozing =0, Slight chance of dozing =1, Moderate chance of dozing =2, High chance of dozing =3
Polysomnography | 1 week after last treatment session.
  • All patients underwent full night attended polysomnography in the sleep laboratory of Mansoura university hospital, Chest department.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansoura City, Eldakahlia, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Attia AAMM, Haggag MA, Ahmed WS, El-Saed A, Saleh MAM, Saleh AM. Dextrose prolotherapy versus low level laser therapy in the treatment of patients with obstructive sleep apnea syndrome; a randomized controlled trial. Sleep Breath. 2025 Aug 12;29(5):272. doi: 10.1007/s11325-025-03428-7. PMID 40794160